CLINICAL TRIAL: NCT01230853
Title: A Randomized, Double-blind, Placebo-controlled, Combined Single Ascending Dose and Multiple Ascending Dose Study to Assess Safety, Tolerability, Immunogenicity, Pharmacodynamic Response, and Pharmacokinetics of Intravenous Infusions of BAN2401 in Subjects With Mild to Moderate Alzheimer?s Disease
Brief Title: A Randomized, Double-blind, Placebo-controlled, Combined Single Ascending Dose and Multiple Ascending Dose Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BAN2401-A001-101
Record Dates: First submitted 2010-10-27; First posted 2010-10-29 (Estimated); Last update posted 2020-11-23 (Actual); Status verified 2013-02

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — lecanemab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Active Comparator: A (Active Comparator)
  Interventions: Drug: Active Comparator: A
- Placebo Comparator A (Placebo Comparator)
  Interventions: Drug: Placebo Comparator A
- Active Comparator: B (Active Comparator)
  Interventions: Drug: Active Comparator B
- Placebo Comparator B (Placebo Comparator)
  Interventions: Drug: Placebo Comparator B

INTERVENTIONS:
Drug: Active Comparator: A — Lecanemab Single Dose Ascending Single intravenous infusions at sequentially ascending doses on Day 1 (dose levels: 0.1, 0.3, 1, 3, 10, and 15 mg/kg)
  Other Names: BAN2401
  Arms: Active Comparator: A
Drug: Placebo Comparator B — Placebo Matching Placebo Infusion
  Arms: Placebo Comparator B
Drug: Active Comparator B — Lecanemab Multiple Dose Ascending Intravenous infusions once every 4 weeks at sequentially ascending doses (dose levels: 0.3, 1, 3, and 10 mg/kg)
  Other Names: BAN2401
  Arms: Active Comparator: B
Drug: Placebo Comparator A — Placebo Matching Placebo Infusion
  Arms: Placebo Comparator A

SUMMARY:
The purpose of this study will be to evaluate the safety and tolerability of lecanemab at sequentially ascending doses in subjects with mild to moderate Alzheimer's disease (AD).

DETAILED DESCRIPTION:
This will be a multicenter, double-blind, randomized, placebo-controlled study in subjects with mild to moderate Alzheimer's disease. The study will comprise separate single dose ascending (SAD) and multiple dose ascending (MAD) parts designed to allow the MAD part to be initiated while the SAD part is ongoing.

ELIGIBILITY:
Inclusion:

1. Clinical diagnosis of probable mild to moderate Alzheimer's disease (AD) by National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association Alzheimer's (NINCDS-ADRDA) criteria.
2. A Mini Mental State Examination (MMSE) score of 16 to 28, inclusive, at Screening. Subjects recruited to the first 2 SAD cohorts should have an MMSE of > 22.
3. Where symptomatic treatment of Alzheimer's disease (AD) is clinically indicated, subjects must be on stable treatment (e.g., with an anticholinesterase inhibitor [AChEI] and/or memantine) for at least 12 weeks prior to the Screening visit.
4. On stable doses of all other prescribed medications for at least 4 weeks prior to the screening visit.

Exclusion:

1. Any neurological condition that could be contributing to cognitive impairment above and beyond that caused by the subject's Alzheimer's disease (AD).
2. Any psychiatric diagnosis or symptoms, e.g hallucinations, major depression, or delusions, that could interfere with assessment of cognition in the subject.
3. History of transient ischemic attack (TIA), stroke, or seizures within 12 months of Screening.
4. Evidence of infection, tumor, stroke or other clinically significant lesions that could indicate a dementia diagnosis other than AD on brain magnetic resonance imaging (MRI) at Screening.
5. Other significant pathological findings on brain MRI at Screening, including but not limited to: more than 3 micro-hemorrhages, single macro-hemorrhage; evidence of vasogenic edema; evidence of cerebral contusion, encephalomalacia, aneurysms, vascular malformations or space occupying lesions.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-08; Primary Completion 2012-10 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Single Ascending Dose (SAD) | baseline to Day 180 post-dose
  To evaluate the safety and tolerability of single intravenous (i.v.) infusions of lecanemab at sequentially ascending doses in subjects with mild to moderate Alzheimer's disease (AD)
Multiple Ascending Dose(MAD) | baseline to Day 264 post-dose
  To evaluate the safety and tolerability of 4 monthly i.v. infusions of lecanemab at sequentially ascending doses in subjects with AD

CONTACTS AND LOCATIONS:
Overall Officials: Eisai Medical Services, Study Director — Eisai Limited
Locations (8):
- United States (8):
  - Garden Grove, California
  - San Francisco, California
  - Orlando, Florida
  - Atlanta, Georgia
  - Indianapolis, Indiana
  - Eatontown, New Jersey
  - Princeton, New Jersey
  - Salt Lake City, Utah

REFERENCES:
- [Derived] Logovinsky V, Satlin A, Lai R, Swanson C, Kaplow J, Osswald G, Basun H, Lannfelt L. Safety and tolerability of BAN2401--a clinical study in Alzheimer's disease with a protofibril selective Abeta antibody. Alzheimers Res Ther. 2016 Apr 6;8(1):14. doi: 10.1186/s13195-016-0181-2. PMID 27048170